CLINICAL TRIAL: NCT02209857
Title: The Symphony Triple A Study: Using Symphony as an Adjunct to Histopathologic Parameters When the Doctor is Ambivalent About the Administration and Type of Adjunctive Systemic Therapy
Brief Title: The Symphony Triple A Study: Using Symphony in Treatment Decisions Concerning Adjuvant Systemic Therapy
Acronym: Symphony
Status: Completed | Type: Observational
Sponsor: Diakonessenhuis, Utrecht (Other)
Collaborators: Agendia (Industry)
Responsible Party: Sponsor
Other Study IDs: DIAK-TrA-20121
Record Dates: First submitted 2014-07-24; First posted 2014-08-06 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Breastcancer; Invasive Breast Carcinoma by Gene Expression Profile
Keywords: Breastcancer; Adjuvant chemotherapy; 70-gene expression profile; MammaPrint

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The tissue specimen for MammaPrint® analysis consists of a tumour block or 10 unstained slides with 5µm section on each slide. The tissue can be shipped as formalin fixed paraffin embedded (FFPE) tissue. For further information: www.agendia.com or www.symphonytripleA.nl.
Oversight: Data Monitoring Committee: No

SUMMARY:
Rationale:

Prediction of prognosis in patients with breast cancer is important to determine the indication for adjuvant chemo-, endocrine- and immunotherapy. Apart from the clinicopathological parameters incorporated into the Adjuvant!Online predictive model, the validated 70-gene signature MammaPrint® is predictive of outcome too. MammaPrint® is advised in the current Dutch CBO guideline (2012) for hormone receptor positive, invasive ductal breast cancer in individual cases when there is 'doubt' about the indication for adjuvant chemotherapy based on traditional prognostic factors. In the present study MammaPrint® is used in this CBO 2012 guideline defined group of patients as an additional test for decision-making for adjuvant chemotherapy.

Objective:

To assess the impact of MammaPrint® on clinical decision making regarding the administration of adjuvant chemotherapy in the CBO 2012 guideline defined group of hormone receptor positive invasive ductal carcinoma patients when there is doubt about the indication for adjuvant chemotherapy based on traditional prognostic factors. The influence of various factors and the impact of MammaPrint® in predefined subgroups will be analyzed too. Data from a national registry regarding adjuvant systemic treatment in patients with similar clinicopathological characteristics in whom MammaPrint® was not used will be obtained to provide a control group.

Hypothesis:

In the group of patients where national guidelines advocate using systemic therapy but doctors are ambivalent in treating patients with adjuvant chemotherapy, it is hypothesized that using MammaPrint® as an additional test will change the indication for adjuvant therapy in a substantial proportion of patients resulting in at least 10% less patients who receive adjuvant chemotherapy. Thus, in the study group at least 10% less patients will receive chemotherapy when compared to a contemporary group of patients with similar clinicopathological characteristics but without using MammaPrint®

Study population:

Hormone receptor positive, invasive ductal breast cancer patients when there is doubt about the indication for adjuvant chemotherapy based on traditional prognostic factors.

Study design:

This is a prospective multicentre impact study.

DETAILED DESCRIPTION:
1. INTRODUCTION AND SCOPE During the last decade treatment guidelines for the administration of adjuvant chemotherapy in patients with breast cancer have changed, today advising chemotherapy in the majority of patients having a >1cm invasive cancer. Prognostic factors used to determine the need for adjuvant chemotherapy are axillary lymph node status, tumour size and grade, patients' age, and HER2 over expression. In addition, HER2 status and ER/PR are also predictive of the effect of particular adjuvant systemic therapies.

   Besides predictive models based on histopathologic factors, gene expression arrays have recognized four different molecular subtypes of breast cancer (Luminal A, Luminal B HER2 +, Luminal B HER2 - and Triple negative). In addition, a number of gene expression profiles have been designed and validated in its capacity to predict the risk of dissemination. One of the gene expression profiles is the 70-gene MammaPrint® signature. The 70-gene MammaPrint® has been validated in different retrospective studies, and in a prospective community-based feasibility study (RASTER). A considerable discrepancy in risk estimations among different clinicopathologic guidelines and MammaPrint was observed. In the RASTER study, addition of MammaPrint to standard clinic-pathological factors led to a change in adjuvant systemic treatment advice in 19% of patients. The 5-year metastases free survival rates for MammaPrint Low Risk (n=219) and High Risk (n=208) patients were 97,0% and 91,7%.

   The recent Dutch CBO guideline (2012) for breast cancer suggests using validated gene expression profiles in individual cases in patients with an invasive ductal carcinoma with positive hormonal receptor when there is doubt about the indication for adjuvant chemotherapy based on the traditional prognostic factors.
2. OBJECTIVES Primary objectives Assess the impact of MammaPrint® on clinical decision making regarding the administration of adjuvant chemotherapy in the CBO 2012 guideline defined group of hormone receptor positive invasive ductal carcinoma patients when there is doubt about the indication for adjuvant chemotherapy based on traditional prognostic factors.

   Secondary objectives
   * To document the influence of primary tumour characteristics (size, Bloom and malignancy grade and Her-2 status) and N-status (N0 vs N1mi) with respect to the (Mammaprint-dependent) decision to give adjuvant chemotherapy in predefined subgroups
   * To address doctor and patient influence on the eventual decision to give adjuvant chemotherapy.

   Hypothesis In the group of patients where contemporary national guidelines advocate using systemic therapy but doctors are ambivalent in treating patients with adjuvant chemotherapy, it is hypothesized that using MammaPrint® as an additional test will change the indication for adjuvant therapy in a substantial proportion of patients resulting in at least 10% less patients who receive adjuvant chemotherapy. Thus, in the study group at least 10% less patients will receive chemotherapy when compared to a contemporary group of patients with similar clinicopathological characteristics but without using MammaPrint®
3. STUDY POPULATION

   Population (base) The study population is the CBO 2012 guideline defined group of hormone receptor positive, invasive ductal breast cancer patients when there is doubt about the indication for adjuvant chemotherapy based on traditional prognostic factors.

   Doubt about the indication for adjuvant chemotherapy based on traditional prognostic factors is an ill-defined criterion. Potential differences in the individual judgement of medical oncologists deciding on adjuvant systemic therapy are conceivable, which will translate in differences in the tendency to use MammaPrint®. Based on the CBO-guideline 2012, we expect that the tendency to use MammaPrint® in small, low-grade tumours as well as in patients with lymph node macrometastases will be relatively low.

   Based on the aforementioned assumptions the expected proportional composition of the study group 'of hormone receptor positive, invasive ductal breast cancer patients when there is doubt about the indication for adjuvant chemotherapy based on traditional prognostic factors' is as follows:

   N0, BR 1, > 2 cm : 10-15% (60-90 patients) N0, BR 2, > 1 cm : 50-60% (300-350 patients) N1mi, grade 1,2 : 15-20% (90-120 patients)

   Her+, N0, <2c, grade I: <5% (<30 patients) NI: <5% (<30 patients) N0, BR 1, 1-2 cm: <5% (<30 patients)

   Control group

   For comparison, data regarding adjuvant chemotherapy in patients in whom no MammaPrint® was used will be obtained from a national registry Netherlands Cancer Registry (NKR) and matched with the MammaPrint® group to date of diagnosis and clinicopathological characteristics. The control group will enable analysis of the impact of Mammaprint on the proportion of patients receiving adjuvant chemotherapy.
4. STUDY DESIGN

This is a prospective multicentre impact study of MammaPrint® on clinical decision making in a predefined group of patients where doctors and patients are ambivalent about adjuvant chemotherapy. MammaPrint® is offered in addition to standard histopathology tests for decision-making regarding adjuvant systemic therapy. The advised adjuvant systemic therapy will be recorded before and after disclosure of the MammaPrint® result.

Logistical planning:

Post-surgery:

1. Every patient is discussed in a multidisciplinary team meeting for further treatment advice. After definitive pathological assessment of tumour size, Bloom and Richardson grade, confirmation of ER/PR- and HER2 status, potential inclusion of a patient is assessed.
2. In the surgical outpatient clinic, patients are seen postoperatively and the histopathological results are discussed. The surgeon informs the patient about the conclusion of the multidisciplinary team and the patient is informed about existing uncertainty of adjuvant treatment and the added value of the MammaPrint. Study information is supplied including an Informed Consent form.
3. The pathologist sends the MammaPrint kit to Agendia for analyses. The attending surgeon and/or research nurse register patients by completing electronic Case Report Form (CRF) 1.
4. MammaPrint® result is emailed to the surgeon, medical oncologist and mammacare nurse within 10 working days.
5. Within two weeks the patient is seen in the outpatient clinic by the oncologist to discuss the result of the MammaPrint®. A final decision concerning adjuvant chemotherapy is made with the patient. CRF 2 is completed by the oncologist.

The study is expected to enrol 600 patients in approximately 25 hospitals in two and a half years. The follow up regarding the advice of adjuvant treatment is estimated to be two months, just after the start of the adjuvant chemotherapy.

5. TISSUE COLLECTION AND 'CLASSIC' HISTOPATHOLOGICAL EXAMINATION

After patients' approval and signed consent forms, samples can be sent to Agendia for MammaPrint® analysis. The tissue specimen for MammaPrint® analysis consists of a tumour block or 10 unstained slides with 5µm section on each slide. The tissue can be shipped as formalin fixed paraffin embedded (FFPE) tissue.

6. STATISTICAL ANALYSIS

Descriptive statistics The primary endpoint is defined as the group of patients who receive adjuvant systemic therapy and will be compared to the proportion of patients who were advised to receive chemotherapy before knowledge of the MammaPrint® result. In addition, using NKR/NBCA data as controls, the absolute difference in the proportion of patients receiving adjuvant chemotherapy is evaluated. This absolute difference is evaluated for the whole group as well as for the three expectedly largest subgroups.

Statistical analysis Baseline characteristics will be summarized by an incidence table. The frequency of chemotherapy + endocrine versus endocrine alone decisions will be addressed before and after receiving the MammaPrint result in the study group. A McNemars test will be performed for the comparison of the two proportions treated (before and after), both expressed as a percentage. When the p- value for this McNemars test is less than 0.05, the conclusion will be that the two proportions indeed differ significantly.

Chi-square tests (binary variables), non-parametric Mann-Whitney test (for continuous variables - 2 groups) and non-parametric Kruskall-Wallis tests (continuous variables - more groups) will be used for the comparison of population characteristics in different subgroups. When the p- values are less than 0.05, the conclusion will be that there is a significant difference between the subgroups for these variables.

The percentage treatment change will be calculated for the whole study group and for the three predefined subgroups. The distribution of MammaPrint test results will be summarized in a frequency table. With a predefined sample size for the whole group (n=600), and a control group consisting of at least 1800 patients the minimal detectable difference in the proportion of patients receiving chemotherapy is 6.6% for the whole group and 9.3% for a subgroup of 300 patients (2-sided alpha 0.05, Power 80). After inclusion of the first 150 patients, additional sample size calculation will be conducted based on the actual proportions of the subgroups.

7. ETHICAL CONSIDERATIONS

Regulation statement This study is conducted according to the principles of the Declaration of Helsinki (version 6, February 2008) and in accordance with the Medical Research Involving Human Subjects Act (WMO) and other legal and regulatory frameworks.

ELIGIBILITY:
Inclusion criteria

* Oestrogen receptor positive, invasive ductal and female breast cancer patients where the benefit of adjuvant chemotherapy is uncertain based on traditional prognostic factors
* Written informed consent
* Patients with multicentric or contralateral disease

Exclusion criteria

* Patients with a previous history of malignancy (in the five years before breast cancer diagnosis), excluding basal cell carcinoma.
* Patients with confirmed distant metastasis.
* Patients who undergo neoadjuvant systemic treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is the CBO 2012 guideline defined group of hormone receptor positive, invasive ductal breast cancer patients when there is doubt about the indication for adjuvant chemotherapy based on traditional prognostic factors. Patients are included and MammaPrint® is determined after complete histological assessment following definitive surgery. The following pathology items have to be recorded: tumour size, grade, ER- and PR- receptor status, Her-2 neu status, and lymph node status. No difference is made in ethnical background or past medical history other than cancer.
Sampling Method: Non-Probability Sample
Enrollment: 660 (Actual)
Dates: Start 2013-01; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Frequency of adjuvant chemotherapy | Within one month after surgery
  We will measure and compare the proportion of patients receiving adjuvant chemotherapy in the group of patients receiving MammaPrint and the group who doesn't receive MammaPrint. In addition we'll record the type of chemotherapy given.

SECONDARY OUTCOMES:
Changes in adjuvant systemic treatment decisions due to MammaPrint use | Within one month after (initial) surgery
  The percentage treatment change will be calculated for the whole study group and for the three predefined subgroups.
Influence of BluePrint and TargetPrint on adjuvant systemic treatment decisions | Within one month after (initial) surgery
  The percentage of adjuvant systemic treatment changes due to the use of BluePrint and/or TargetPrint for the whole studygroup, and the various subgroups will be calculated.
Clinical utility of MammaPrint in multicentric/contralateral disease. | Within one month after (initial) surgery
  Of patients included in the Symphony Triple A study with multicentric or contralateral breast cancer two tissue samples will be collected and a MammaPrint will be performed on both samples. In this subgroup of patients, MammaPrint, BluePrint and TargetPrint results of both tumors will be compared to evaluate the clinical utility of MammaPrint in multicentric and contralateral disease.
Concordance of TargetPrint results with locally assessed ICH/FISH ER, PR and Her2 results | Within one month after (initial) surgery
  The concordance between the ER, PR and Her2 results as assessed by the TargetPrint and local ICH/FISH techniques will be assessed.
Comparison of clinical subtype with BluePrint molecular subtype | Within one month after (initial) surgery
  Based on the ER, PR and Her2 results as assessed by local pathologist patients can be categorized in clinical molecular subtypes. Concordance between these clinical subtypes and the molecular subtype as assessed by the BluePrint will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Thijs van Dalen, Dr, Principal Investigator — Diakonessenhuis Utrecht, The Netherlands
Locations (34):
- Netherlands (34):
  - Whilhelmina ziekenhuis, Assen, Drenthe
  - Medisch Centrum Zuiderzee, Lelystad, Flevoland
  - Gelre ziekenhuis, Apeldoorn, Gelderland
  - Rijnstate, Arnhem, Gelderland
  - Gederse Vallei, Ede, Gelderland
  - Sint Jansdal, Harderwijk, Gelderland
  - Ziekenhuis Rivierenland, Tiel, Gelderland
  - Gelre ziekenhuis, Zutphen, Gelderland
  - Jeroen Bosch ziekenhuis, 's-Hertogenbosch, North Brabant
  - Medisch Centrum Alkmaar, Alkmaar, North Holland
  - Boven IJ ziekenhuis, Amsterdam, North Holland
  - Onze Lieve Vrouwe Gasthuis, Amsterdam, North Holland
  - Gemini ziekenhuis, Den Helder, North Holland
  - Kennemer Gasthuis, Haarlem, North Holland
  - Spaarne ziekenhuis, Hoofddorp, North Holland
  - Westfriesgasthuis, Hoorn, North Holland
  - Waterland ziekenhuis, Purmerend, North Holland
  - Vlietland ziekenhuis, Schiedam, North Holland
  - Zaans medisch centrum, Zaandam, North Holland
  - Deventer ziekenhuis, Deventer, Overijssel
  - Ropcke Zweers ziekenhuis, Hardenberg, Overijssel
  - Isale klinieken, Zwolle, Overijssel
  - Nij Smellinghe ziekenhuis, Drachten, Provincie Friesland
  - Tjongerschans, Heerenveen, Provincie Friesland
  - Antoniusziekenhuis, Sneek, Provincie Friesland
  - Martini ziekenhuis, Groningen, Provincie Groningen
  - IJsselland ziekenhuis, Capelle aan den IJssel, South Holland
  - Sint Fransiscus gasthuis, Rotterdam, South Holland
  - Lange Land ziekenhuis, Zoetermeer, South Holland
  - Alexander Monro ziekenhuis, Bilthoven, Utrecht
  - Ter Gooi ziekenhuis, Hilversum, Utrecht
  - Sint Antoniusziekenhuis, Nieuwegein, Utrecht
  - Diakonessenziekenhuis, Utrecht, Utrecht
  - Zuwe Hofpoort ziekenhuis, Woerden, Utrecht

REFERENCES:
- [Background] Ravdin PM, Siminoff LA, Davis GJ, Mercer MB, Hewlett J, Gerson N, Parker HL. Computer program to assist in making decisions about adjuvant therapy for women with early breast cancer. J Clin Oncol. 2001 Feb 15;19(4):980-91. doi: 10.1200/JCO.2001.19.4.980. PMID 11181660
- [Background] Perou CM, Sorlie T, Eisen MB, van de Rijn M, Jeffrey SS, Rees CA, Pollack JR, Ross DT, Johnsen H, Akslen LA, Fluge O, Pergamenschikov A, Williams C, Zhu SX, Lonning PE, Borresen-Dale AL, Brown PO, Botstein D. Molecular portraits of human breast tumours. Nature. 2000 Aug 17;406(6797):747-52. doi: 10.1038/35021093. PMID 10963602
- [Background] van de Vijver MJ, He YD, van't Veer LJ, Dai H, Hart AA, Voskuil DW, Schreiber GJ, Peterse JL, Roberts C, Marton MJ, Parrish M, Atsma D, Witteveen A, Glas A, Delahaye L, van der Velde T, Bartelink H, Rodenhuis S, Rutgers ET, Friend SH, Bernards R. A gene-expression signature as a predictor of survival in breast cancer. N Engl J Med. 2002 Dec 19;347(25):1999-2009. doi: 10.1056/NEJMoa021967. PMID 12490681
- [Background] van 't Veer LJ, Dai H, van de Vijver MJ, He YD, Hart AA, Mao M, Peterse HL, van der Kooy K, Marton MJ, Witteveen AT, Schreiber GJ, Kerkhoven RM, Roberts C, Linsley PS, Bernards R, Friend SH. Gene expression profiling predicts clinical outcome of breast cancer. Nature. 2002 Jan 31;415(6871):530-6. doi: 10.1038/415530a. PMID 11823860
- [Background] Buyse M, Loi S, van't Veer L, Viale G, Delorenzi M, Glas AM, d'Assignies MS, Bergh J, Lidereau R, Ellis P, Harris A, Bogaerts J, Therasse P, Floore A, Amakrane M, Piette F, Rutgers E, Sotiriou C, Cardoso F, Piccart MJ; TRANSBIG Consortium. Validation and clinical utility of a 70-gene prognostic signature for women with node-negative breast cancer. J Natl Cancer Inst. 2006 Sep 6;98(17):1183-92. doi: 10.1093/jnci/djj329. PMID 16954471
- [Background] Bueno-de-Mesquita JM, Linn SC, Keijzer R, Wesseling J, Nuyten DS, van Krimpen C, Meijers C, de Graaf PW, Bos MM, Hart AA, Rutgers EJ, Peterse JL, Halfwerk H, de Groot R, Pronk A, Floore AN, Glas AM, Van't Veer LJ, van de Vijver MJ. Validation of 70-gene prognosis signature in node-negative breast cancer. Breast Cancer Res Treat. 2009 Oct;117(3):483-95. doi: 10.1007/s10549-008-0191-2. Epub 2008 Sep 26. PMID 18819002
- [Background] Mook S, Schmidt MK, Viale G, Pruneri G, Eekhout I, Floore A, Glas AM, Bogaerts J, Cardoso F, Piccart-Gebhart MJ, Rutgers ET, Van't Veer LJ; TRANSBIG Consortium. The 70-gene prognosis-signature predicts disease outcome in breast cancer patients with 1-3 positive lymph nodes in an independent validation study. Breast Cancer Res Treat. 2009 Jul;116(2):295-302. doi: 10.1007/s10549-008-0130-2. Epub 2008 Jul 27. PMID 18661261
- [Background] Knauer M, Mook S, Rutgers EJ, Bender RA, Hauptmann M, van de Vijver MJ, Koornstra RH, Bueno-de-Mesquita JM, Linn SC, van 't Veer LJ. The predictive value of the 70-gene signature for adjuvant chemotherapy in early breast cancer. Breast Cancer Res Treat. 2010 Apr;120(3):655-61. doi: 10.1007/s10549-010-0814-2. Epub 2010 Mar 5. PMID 20204499
- [Background] Mook S, Schmidt MK, Weigelt B, Kreike B, Eekhout I, van de Vijver MJ, Glas AM, Floore A, Rutgers EJT, van 't Veer LJ. The 70-gene prognosis signature predicts early metastasis in breast cancer patients between 55 and 70 years of age. Ann Oncol. 2010 Apr;21(4):717-722. doi: 10.1093/annonc/mdp388. Epub 2009 Oct 13. PMID 19825882
- [Background] Mook S, Knauer M, Bueno-de-Mesquita JM, Retel VP, Wesseling J, Linn SC, Van't Veer LJ, Rutgers EJ. Metastatic potential of T1 breast cancer can be predicted by the 70-gene MammaPrint signature. Ann Surg Oncol. 2010 May;17(5):1406-13. doi: 10.1245/s10434-009-0902-x. Epub 2010 Jan 22. PMID 20094918
- [Background] Bueno-de-Mesquita JM, van Harten WH, Retel VP, van 't Veer LJ, van Dam FS, Karsenberg K, Douma KF, van Tinteren H, Peterse JL, Wesseling J, Wu TS, Atsma D, Rutgers EJ, Brink G, Floore AN, Glas AM, Roumen RM, Bellot FE, van Krimpen C, Rodenhuis S, van de Vijver MJ, Linn SC. Use of 70-gene signature to predict prognosis of patients with node-negative breast cancer: a prospective community-based feasibility study (RASTER). Lancet Oncol. 2007 Dec;8(12):1079-1087. doi: 10.1016/S1470-2045(07)70346-7. Epub 2007 Nov 26. PMID 18042430
- [Background] Drukker CA, Bueno-de-Mesquita JM, Retel VP, van Harten WH, van Tinteren H, Wesseling J, Roumen RM, Knauer M, van 't Veer LJ, Sonke GS, Rutgers EJ, van de Vijver MJ, Linn SC. A prospective evaluation of a breast cancer prognosis signature in the observational RASTER study. Int J Cancer. 2013 Aug 15;133(4):929-36. doi: 10.1002/ijc.28082. Epub 2013 Mar 4. PMID 23371464
- See also: Information concerning the MammaPrint 70-gene expression profile — http://www.agendia.com//
- See also: Current Dutch national guideline breast cancer — http://www.oncoline.nl/mammacarcinoom